CLINICAL TRIAL: NCT01938170
Title: A Pilot Study to Assess the Acceptability, Tolerability, and Feasibility of Home Intranasal Administration of FluMist® by a Trained Primary Caregiver to Healthy Family Members 2 Through 17 Years of Age
Brief Title: Home Administration of FluMist by Parents/Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of North Carolina (Other); MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-2769
Record Dates: First submitted 2013-08-23; First posted 2013-09-10 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FluMist (Experimental): Subjects receiving vaccine at home
  Interventions: Biological: FluMist

INTERVENTIONS:
Biological: FluMist — Subjects receiving Flumist vaccine

SUMMARY:
This study will examine the feasibility of having parents and caregivers administer FluMist live intranasal vaccine to their children at home outside the traditional medical environment and without the involvement of medical personnel.

The study will recruit patients and families that are already eligible to receive the FluMist vaccine. After consent is obtained and vaccine is given to the family, they will go home to administer vaccine to other members within 24 hours. Telephone follow up within 48 hours will confirm that vaccine was given successfully and within 9-12 days to assess patient preferences for giving vaccine at home and if there were any adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. The primary caregiver must be 18 years of age or older and willing to give written informed consent for study participation
2. The primary caregiver must be the parent or legal guardian of all the children in living in the household
3. All the children in the household who are 2 through 17 years of age must receive their primary care in the clinic
4. All the children in the household who are 2 through 17 years of age must have private insurance that will provide for the cost of influenza vaccination
5. There must be at least one member of the household who is 2 through 17 years of age, presenting for care in the clinic, eligible to receive Live Attenuated Influenza Vaccine (LAIV) and whose primary care giver is willing to administer LAIV to them in the clinic with supervision
6. There must be at least one family member of the household who is 2 through 17 years of age, not presenting for care in the clinic, eligible to receive LAIV and whose primary care giver is willing to administer LAIV to them in the in-home setting
7. There must be a working refrigerator in the household
8. The primary caregiver must have a working telephone number and be willing to be contacted for study follow-up by telephone or e-mail
9. The primary caregiver is available for the entire study period - 12 days following the last dose of LAIV to be administered to a child
10. The primary caregiver must agree to complete a 30 minute post vaccination assessment and an 8 day diary following vaccination for each child receiving LAIV.

Exclusion Criteria:

1. Children in the family receive vaccine through Vaccines for Children program

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Jhaveri, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Jhaveri R, Allyne K. A Feasibility Trial of Home Administration of Intranasal Vaccine by Parents to Eligible Children. Clin Ther. 2017 Jan;39(1):204-211.e4. doi: 10.1016/j.clinthera.2016.11.018. Epub 2016 Dec 7. PMID 27938896

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10/2014-1/2015
Period: Overall Study
Arm/Group | FluMist
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FluMist
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Reported Successful Home Vaccination With no Adverse Events
Description: We will assess the tolerability of giving the FluMist nasal vaccine at home by parents/caregivers to their children by performing telephone survey follow up. We will ask parents at both 24-48 hours and at 9-12 days after study visit and enrollment about any difficulties in giving FluMist at home and any adverse events encountered when giving FluMist at home.
Time Frame: 0-12 days
Measure: Number; unit: participants
Arm/Group | FluMist
Number analyzed (Participants) | 41
participants | 41

2. Secondary Outcome: Number of Subjects That Reported Ability to Successfully Administer FluMist Vaccine at Home
Description: This study will also assess the feasibility of having parents/caregivers administer Flumist vaccine outside a traditional medical environment and without the direct participation of medical personnel. We will ask parents by telephone survey at both 24-48 hours and at 9-12 days after study visit and enrollment about any difficulties in giving FluMist at home, about maintaining temperature and conditions proper for vaccine storage until administration. We will also ask about ease of vaccine disposal and about child preferences for receiving vaccine at home compared to at a dedicated medical visit.
Time Frame: 0-12 days
Measure: Number; unit: participants
Arm/Group | FluMist
Number analyzed (Participants) | 41
participants | 41

ADVERSE EVENTS:
Arm/Group | FluMist
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 10/41
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FluMist (N=41)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Fatigue (General disorders) | 2 (2)
Sore Throat (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Vomiting (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No